CLINICAL TRIAL: NCT01352338
Title: A Phase 1 and Phase 2 Study of Lenalidomide (Revlimid) in Combination With Cyclophosphamide (Endoxan) and Prednison (REP) in Relapsed/Refractory Multiple Myeloma
Brief Title: Revlimid, Endoxan, Prednison Evaluation After Prior Revlimid Treatment (REPEAT)
Acronym: REPEAT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Principal Investigator, I.S. Nijhof, Drs, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RV-MM-PI-0630
Record Dates: First submitted 2011-04-13; First posted 2011-05-11 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Multiple Myeloma
Keywords: REPEAT; multiple myeloma; revlimid; lenalidomide; cyclophosphamide; endoxan; prednisone; lenalidomide refractory
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; Cyclophosphamide; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- lenalidomide, endoxan, prednisone (Experimental): lenalidomide 25mg, oral therapy, once a day, 4 weeks cycles. Lenalidomide is used 3 of the 4 weeks.
  Lenalidomide is combined with endoxan and prednisone
  Interventions: Drug: Lenalidomide, endoxan, prednisone

INTERVENTIONS:
Drug: Lenalidomide, endoxan, prednisone — dose-finding
  Other Names: revlimid combined with endoxan and prednisone
Drug: lenalidomide, endoxan, prednisone — oral therapy with lenalidomide 25mg a day during 3 of 4 week cycles. Number of Cycles: until progression or unacceptable toxicity develops.
  Other Names: revlimid combined with cyclophosphamide and prednisone

SUMMARY:
Study Phase: phase 1 and phase 2

Objective: Evaluation of the effect of lenalidomide, cyclophophamide and prednisone (REP) in patients with relapsed multiple myeloma previously treated with lenalidomide

Study design: prospective, multicenter, non-randomized

DETAILED DESCRIPTION:
The REPEAT-study is a prospective, multicenter, non-randomized phase 1 and phase 2 study in which we evaluate the effect of lenalidomide, cyclophosphamide and prednisone (REP-therapy) in patients with relapsed multiple myeloma, previously treated with lenalidomide and refractory to lenalidomide monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* salmon & Durie stage II/III A or B
* previous lenalidomide refractory disease
* patient commits to pregnancy prevention programme

Exclusion Criteria:

* non-secretory myeloma
* known hypersensitivity to lenalidomide
* inadequate marrow reserve

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2011-08; Primary Completion 2014-11 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Phase 1 Revlimid, Endoxan, Prednisone Evaluation After prior revlimid Treatment (REPEAT) | 29 days after start of treatment cycle 1
  To determine the maximum tolerated dose (MTD) and recommended phase 2 dose level (RDL) of lenalidomide administered during 21 days of a 4 weeks cycle, combined with continuous cyclophosphamide and prednisone

SECONDARY OUTCOMES:
phase 1 part of the study Revlimid, Endoxan, Prednison Evaluation After prior revlimid Treatment (REPEAT) | 29 days after start of treatment cycle 1
  number of participants with adverse events
phase 2 part of the study Revlimid, Endoxan, Prednison Evaluation After prior revlimid Treatment (REPEAT) | 28 days
  - to evaluate progression-free survival
phase 2 part of the study Revlimid, Endoxan, Prednison Evaluation After prior revlimid Treatment (REPEAT) | 28 days
  - to evaluate overall survival
phase 2 part of the study Revlimid, Endoxan, Prednison Evaluation After prior revlimid Treatment (REPEAT) | 28 days
  - to evaluate the immunomodulatory effects of lenalidomide by using flow cytometric and cytokine analysis

CONTACTS AND LOCATIONS:
Overall Officials: Dr. N.C.W.J. Donk, van de, MD PhD, Principal Investigator — UMC Utrecht
Locations (3):
- Netherlands (3):
  - Antonius Ziekenhuis Nieuwegein, Nieuwegein, Utrecht
  - UMC Utrecht, Utrecht, Utrecht
  - VU Medical Center, Amsterdam

REFERENCES:
- [Derived] Nijhof IS, Franssen LE, Levin MD, Bos GMJ, Broijl A, Klein SK, Koene HR, Bloem AC, Beeker A, Faber LM, van der Spek E, Ypma PF, Raymakers R, van Spronsen DJ, Westerweel PE, Oostvogels R, van Velzen J, van Kessel B, Mutis T, Sonneveld P, Zweegman S, Lokhorst HM, van de Donk NWCJ. Phase 1/2 study of lenalidomide combined with low-dose cyclophosphamide and prednisone in lenalidomide-refractory multiple myeloma. Blood. 2016 Nov 10;128(19):2297-2306. doi: 10.1182/blood-2016-07-729236. Epub 2016 Sep 19. PMID 27647864